CLINICAL TRIAL: NCT05550701
Title: Prognostic Impact of Increased Lymph Node Yield in Colorectal Cancer Patients With Synchronous Distant Metastasis: a Population-based Study of the US Database and a Chinese Registry
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Harbin Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Shuai Jiao, doctor, The Second Affiliated Hospital of Harbin Medical University
Other Study IDs: SZSM201911012
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer Stage IV; Lymph Node Yield
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SEER database: Data on CRC patients with synchronous liver metastasis (LM) were derived from the US Surveillance, Epidemiology, and End Results (SEER) between January 2010 and December 2017.
  Interventions: Other: lymph node yield
- Chinese cohort: Data on CRC patients with synchronous liver metastasis (LM) were derived from two Chinese tertiary centers: The Second Affiliated Hospital of Harbin Medical University and National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College between January 2010 and December 2017.
  Interventions: Other: lymph node yield

INTERVENTIONS:
Other: lymph node yield — We recorded the number of lymph nodes dissected during surgery in patients with colorectal cancer

SUMMARY:
The National Quality Forum has endorsed at least 12 lymph node yield (LNY) as a surgical quality indicator in colorectal cancer (CRC), but the prognostic value of adequate lymphadenectomy has rarely been investigated for CRC patients with distant metastatic disease.

DETAILED DESCRIPTION:
Data on CRC patients with synchronous liver metastasis (LM) were derived from the US Surveillance, Epidemiology, and End Results (SEER) and a Chinese registry (from two Chinese tertiary centers: The Second Affiliated Hospital of Harbin Medical University and National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College) between January 2010 and December 2017. Individual level data on patients with incident CRC were consecutively collected in both registries. The primary tumor site was divided into three subsites according to International Classification of Diseases for Oncology (ICD-O-3) topography codes: proximal colon (C18.0, C18.1, C18.2, C18.3 and C18.4), distal colon (C18.5, C18.6, C18.7) and rectum (C19.9 and C20.9). The synchronous LM were identified by imaging or histopathological examinations. Synchronous LM refers to liver lesions found within 6 months after the diagnosis of primary CRC. Patients were excluded if they did not undergo surgery for CRC, did not have data on number of LNs retrieved and their survival status was unknown.

ELIGIBILITY:
Inclusion Criteria:

* Data on CRC patients with synchronous liver metastasis (LM) undergo surgery for CRC, have data on number of LNs retrieved and their survival status was known

Exclusion Criteria:

* Patients were excluded if they did not undergo surgery for CRC, did not have data on number of LNs retrieved and their survival status was unknown

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the US Surveillance, Epidemiology, and End Results (SEER) and a Chinese registry (from two Chinese tertiary centers: The Second Affiliated Hospital of Harbin Medical University and National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College) between January 2010 and December 2017
Sampling Method: Probability Sample
Enrollment: 4575 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
cancer specific survival | 2010.01-2017.12
  The primary outcome was cancer specific survival (CSS), which was defined as the time interval from the synchronous LM diagnosis until cancer specific death or the end of follow-up in Chinese registry, and the CSS was defined using the SEER cause-of-death codes in SEER registry

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics and ethics of the Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
The data involves the relevant personal privacy information of the patient

REFERENCES:
- [Background] Doll KM, Rademaker A, Sosa JA. Practical Guide to Surgical Data Sets: Surveillance, Epidemiology, and End Results (SEER) Database. JAMA Surg. 2018 Jun 1;153(6):588-589. doi: 10.1001/jamasurg.2018.0501. No abstract available. PMID 29617544
- [Background] Thomas L, Li F, Pencina M. Using Propensity Score Methods to Create Target Populations in Observational Clinical Research. JAMA. 2020 Feb 4;323(5):466-467. doi: 10.1001/jama.2019.21558. No abstract available. PMID 31922529
- [Derived] Jiao S, Guan X, Zhang W, Wei R, Wang G, Wang X. Prognostic impact of increased lymph node yield in colorectal cancer patients with synchronous liver metastasis: a population-based retrospective study of the US database and a Chinese registry. Int J Surg. 2023 Jul 1;109(7):1932-1940. doi: 10.1097/JS9.0000000000000244. PMID 37037584